CLINICAL TRIAL: NCT04046835
Title: The Effect of Patient Position on the External Haller Index Value Among Patients With Pectus Excavatum
Acronym: POSITION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ20190106
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Pectus Excavatum
Keywords: Three-dimensional optical surface scanning; Patient position
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pectus excavatum is the most common anterior chest wall deformity, affecting up to 1:400 of newborns. The current gold standard to quantify the extent of deformity is by calculating the Haller Index based on a Computed Tomography (CT)-scan. However, as such scans inescapably imply exposure to ionizing radiation, novel imaging techniques have been investigated. Three-dimensional optical surface scanning is a promising new technique to acquire the trunks' three-dimensional (3D) surface topography. Based on this 3D scan, one is able to calculate the external Haller Index that is known to highly correlate with the conventional gold standard Haller Index that is based on internal measures. Both the conventional and external Haller Index are known to be affected by the respiratory phase in which the scan is acquired, however, what is the effect of patient position on the external Haller Index, and if affected, how should one correct for this phenomenon? To investigate this, a retrospective single-centre pilot study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received a three-dimensional optical surface scan to quantify their pectus deformity

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that received a three-dimensional optical surface scan to quatify their pectus deformity utilizing the external Haller Index. Patients were retrospectively recruited from the 3DPECTUS study (METCZ20190048; NCT03926078).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Patient position | 5 months
  The effect of patient position on the value of the external Haller Index, based on 3D scans.

SECONDARY OUTCOMES:
Manual versus automatic alignment of patient position | 5 months
  If there is a significant effect of patient position on the external Haller Index, the ideal correction method is investigated (manual alignment versus automatic, computer-based alignment)

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands